CLINICAL TRIAL: NCT05346718
Title: Determination of Threshold Concentrations for Ragweed and Birch Pollen in Sensitized Patients with Seasonal Allergic Rhinitis in an Allergen Challenge Chamber and in Vitro
Brief Title: Threshold Concentrations for Ragweed and Birch Pollen in Seasonal Allergic Rhinitis
Acronym: UBAMBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jens Hohlfeld, MD, Division Director of Airway Research, Fraunhofer-Institute of Toxicology and Experimental Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-08 UBAMBI
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Allergic Rhinitis; Seasonal Allergic Rhinitis; Ragweed Allergy; Birch Pollen Allergy
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — ragweed pollen

STUDY DESIGN:
Intervention Model Description: The study design is mixed. Participants are randomized to the sequence of the placebo and first pollen concentration (cross over). Then they are exposed as a single group in all following allergen challenges.
Who Masked: Participant
Masking Description: Participants are blinded to the pollen concentration of each allergen challenge, including placebo exposure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A: Exposure to no pollen (placebo), then to first pollen concentration (Experimental): Participants are first exposed to no pollen, then challenged with the first pollen concentration, and finally all following concentrations.
  Interventions: Other: Ragweed pollen, birch pollen, clean air (placebo)
- Sequence B: Exposure to first pollen concentration, then to no pollen (placebo) (Experimental): Participants are first challenged with the first pollen concentration, then with no pollen, and finally with all following concentrations.
  Interventions: Other: Ragweed pollen, birch pollen, clean air (placebo)

INTERVENTIONS:
Other: Ragweed pollen, birch pollen, clean air (placebo) — Participants are exposed for 4 hours in the Fraunhofer Allergen Challenge Chamber with varying pollen concentrations of ragweed or birch pollen and once with clean air, serving as a placebo exposure.

SUMMARY:
The ragweed Ambrosia artemisiifolia is spreading in northern Europe due to climate change. The pollen are considered highly allergenic and might trigger allergy symptoms at much lower concentrations than e.g. grass or birch pollen. This study aims to determine threshold concentrations for ragweed and birch pollen in patients with seasonal allergic rhinitis. Participants will be exposed in an allergen challenge chamber that was technically modified to maintain very low and stable pollen concentrations for several hours. The study design is adaptive, where the pollen concentrations are escalated or de-escalated based on interim analysis of resulting allergic symptoms.

DETAILED DESCRIPTION:
Ambrosia artemisiifolia (hereafter briefly referred to as ragweed) is an anemophilous herb of the Asteraceae family that probably originated in desert areas of the USA. The plant was introduced to Europe through trade and spread as a successful neophyte during the 20th century. Although conditions are not ideal for ragweed in northern and central Europe, when the plant prefers dry, sandy soils, climate change may be a significant contributor to its spread. The pollen is considered highly allergenic, so it is possible that lower pollen concentrations are sufficient to trigger allergy symptoms compared to native grass or birch pollen. Together with its ability to spread invasively and its tolerance to harmful factors, ragweed is therefore considered a health hazard.

Determining threshold concentrations for various aeroallergens has been attempted many times in published literature. In fact, first experiments have been reported since the 1960s. However, obtaining comparable results prove difficult due to a plethora of methods, outcome measures and choices in study population. Basically, threshold concentration could be assessed by target organ specific allergen challenge, field study and allergen chamber challenge - each of which has its own benefits and drawbacks.

To date, allergen challenge chambers have been used primarily for proof-of-concept studies with antiallergic agents. Technically, the chambers are designed to maintain high pollen concentrations, which should induce symptoms in all sensitized subjects, at a constant level for hours in order to be able to determine the maximum possible effect size of the investigated therapeutic intervention. Metering and monitoring of pollen to maintain stable concentrations present technical challenges for deploying pollen concentrations in the double-digit range. Fraunhofer ITEM has successfully established low concentration pollen exposures, so that allergic patients can be titrated to effect. The pollen concentration will be escalated or de-escalated according to a pre-defined algorithm, based on interim data analysis. Eventually, a concentration range for ragweed and birch pollen can be determined that induces allergic symptoms with clinical and statistical significance.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent.
2. Male and female subjects, aged 18-65 years. Women will be considered for inclusion if they are:

   1. Not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing.
   2. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit).
   3. Of childbearing potential and using a highly effective birth control during the entire study as described in section 8.2.
3. Body mass index between 18 and 35 kg/m2.
4. History of seasonal allergic rhinitis to ragweed (July to September) or birch pollen (March to May).
5. Positive skin prick test response (positive wheal diameter reaction of ≥ 3mm) for Ambrosia artemisiifolia or Betula pendula at screening or within 12 months prior to screening visit.
6. Subject has a serum specific IgE level (≥ 0.7 kU/L) to Ambrosia artemisiifolia or Betula pendula at screening or within the past 12 months (record required).
7. Normal lung function (FEV1 ≥ 80% pred. and FEV1/FVC ≥ LLN) at screening. If subject fails to meet criteria, assessment may be repeated 2 additional times.
8. TNSS of 0 prior to entering the ACC at all exposures.
9. Mild to moderate level of rhinitis symptoms in the screening challenge to ragweed or birch, defined as a mean TNSS between 1 to 8 after the 4-hour ACC and a TNSS continuously > 0 after 40 minutes.

Exclusion Criteria:

1. Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urinalysis, vital signs, lung function or ECG at screening visit , which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or may influence the results of the study, or the subject's ability to participate in the study.
2. Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
3. Subjects with concomitant allergies to seasonal aeroallergens (i.e., grass, trees, weeds, rye; defined as IgE ≥ 3.5 kU/L within the last 12 months prior to screening) which are anticipated to be or become active during study participation.
4. Subjects with a symptomatic concomitant allergy to an animal dander being exposed during study participation.
5. Subjects with a symptomatic house dust mite allergy.
6. Symptoms of a respiratory tract infection within 3 days prior to screening. Subjects may be re-screened if they have been asymptomatic for at least 3 days.
7. Asthma requiring more than Step 1 medication according to GINA guidelines (Global Initiative for Asthma Management and Prevention, 2021). Asthmatic subjects taking ICS plus long-acting bronchodilator as needed according to Step 1 must to be switched to salbutamol as needed during study participation.
8. Intake of prohibited medication (refer to Section 9.2).
9. Smokers who are unable to refrain from smoking within 1 hr prior to and during visits.
10. Anatomical nasal abnormalities, pronounced nasal septum deviation or nasal polyps blocking nasal air flow on examination or recent nasal surgery.
11. Participation in a clinical trial with a medicinal product or medical device 30 days prior to Visit 1.
12. History of drug or alcohol abuse in the past 12 months.
13. Specific Immunotherapy (SIT) against birch or ragweed within 5 years prior to the study.
14. Risk of non-compliance with study procedures.
15. Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Threshold concentrations for ragweed and birch pollen | Day 1, Day 7, Day 14, Day 21, Day 28 (at least 3 exposure visits, maximum 5 exposure visits)
  Changes in mean Total Nasal Symptom Score (TNSS) of 140 to 240 minutes, nasal secretion, and peak nasal inspiratory flow (PNIF) after challenge with ragweed and birch pollen compared to placebo challenge

SECONDARY OUTCOMES:
Determining allergenic potency of ragweed compared to birch pollen | Day 1, Day 7, Day 14, Day 21, Day 28 (at least 3 exposure visits, maximum 5 exposure visits)
  Mean TNSS of 140 to 240 minutes after challenge with ragweed pollen compared to birch pollen
Basophil activation under varying pollen concentrations in vitro | Screening visit
  CD63 expression (%) on whole blood basophils after stimulation with increasing concentrations of ragweed or birch pollen compared to negative control
Neutrophil migration under varying pollen concentrations in vitro | Screening visit
  Neutrophil migration (% above basal migration) towards increasing concentrations of ragweed or birch pollen compared to negative control

OTHER OUTCOMES:
Measuring changes in fractioned exhaled nitric oxide before and after allergen challenges | Day 1, Day 7, Day 14, Day 21, Day 28 (at least 3 exposure visits, maximum 5 exposure visits)
  Changes in nasal fractionated exhaled nitric oxide (FeNO) after challenge with ragweed and birch pollen compared to pre challenge nasal FeNO and placebo challenge
Measuring changes in proinflammatory biomarkers before and after allergen challenges | Day 1, Day 2; Day 7, Day 8; Day 14, Day 15; Day 21, 22; Day 28, 29 (at least 3 exposure visits, maximum 5 exposure visits)
  Changes in inflammatory biomarkers such as histamine, eotaxin, IL-4, IL-5, IL-6, IL-13, TNF-α and MIP-1β after challenge with ragweed and birch pollen compared to pre challenge and placebo measurements from nasal filter papers
Measuring changes in proinflammatory cells before and after allergen challenges | Day 1, Day 2; Day 7, Day 8; Day 14, Day 15; Day 21, 22; Day 28, 29 (at least 3 exposure visits, maximum 5 exposure visits)
  Changes in concentration of eosinophil and neutrophil granulocytes, macrophages, lymphocytes and monocytes after challenge with increasing cumulative exposures to ragweed and birch pollen compared to pre challenge and placebo measurements from nasal lavage
Measuring changes in basophil surface antigen expression under varying pollen concentrations in vitro | Screening visit
  CD63 (%) and CD203c (median fluorescence intensity) expression on whole blood basophils after stimulation with increasing concentrations of ragweed or birch major allergens compared to negative control
Measrung neutrophil migration under varying pollen major allergens concentrations in vitro | Screening visit
  Neutrophil migration (% above basal migration) towards increasing concentrations of ragweed or birch major allergens compared to negative control

CONTACTS AND LOCATIONS:
Overall Officials: Jens M Hohlfeld, Prof. Dr., Principal Investigator — Fraunhofer Institute for Toxicology and Experimental Medicine ITEM
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine, Hanover, Lower Saxony, Germany

REFERENCES:
- [Background] Gaudeul M, Giraud T, Kiss L, Shykoff JA. Nuclear and chloroplast microsatellites show multiple introductions in the worldwide invasion history of common ragweed, Ambrosia artemisiifolia. PLoS One. 2011 Mar 10;6(3):e17658. doi: 10.1371/journal.pone.0017658. PMID 21423697
- [Background] Buters J, Alberternst B, Nawrath S, Wimmer M, Traidl-Hoffmann C, Starfinger U, Behrendt H, Schmidt-Weber C, Bergmann KC. Ambrosia artemisiifolia (ragweed) in Germany - current presence, allergological relevance and containment procedures. Allergo J Int. 2015;24:108-120. doi: 10.1007/s40629-015-0060-6. Epub 2015 Jul 11. PMID 27226949
- See also: Participant recruitment site of Fraunhofer ITEM for this study — https://www.probanden.fraunhofer.de/de/proband-werden/allergien/studie-ubambi.html